CLINICAL TRIAL: NCT04718493
Title: Endoscopic Stenting in Crohn Related Strictures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Per Hedenström, Dr, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Project database VGR 95381
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Intestinal Strictures Related to Crohn´s Disease
MeSH Terms: interventions — Self Expandable Metallic Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stent (Experimental)
  Interventions: Procedure: Self-expandable metal stent
- Dilatation (Active Comparator)
  Interventions: Procedure: Balloon dilatation

INTERVENTIONS:
Procedure: Self-expandable metal stent — Endoscopic stenting of intestinal stricture related to Crohn´s disease
  Arms: Stent
Procedure: Balloon dilatation — Endoscopic balloon dilatation of intestinal stricture related to Crohn´s disease
  Arms: Dilatation

SUMMARY:
Prospective, randomized-controlled trial comparing self-expandable metal stent versus ballon dialtation only for the endoscopic treatment of benign strictures related to Crohn´s disease.

ELIGIBILITY:
Inclusion Criteria:

* Benign high-grade Crohn stricture

Exclusion Criteria:

* Unwillingness to participate
* Planned surgery
* High risk for bleeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Technical success rate | Peroperative
Adverse event rate | Within 7 days

SECONDARY OUTCOMES:
Clinical success rate | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Per-Ove Stotzer, Ass Prof, Principal Investigator — Sahlgrenska University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hedenstrom P, Stotzer PO. Endoscopic treatment of Crohn-related strictures with a self-expandable stent compared with balloon dilation: a prospective, randomised, controlled study. BMJ Open Gastroenterol. 2021 Mar;8(1):e000612. doi: 10.1136/bmjgast-2021-000612. PMID 33722805